CLINICAL TRIAL: NCT06131840
Title: An Open-label Phase 1 Study to Investigate PF-08046050 (SGN-CEACAM5C) in Adults With Advanced Solid Tumors
Brief Title: A Study of SGN-CEACAM5C in Adults With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Seagen, a wholly owned subsidiary of Pfizer (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Organization: Seagen Inc. (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SGNCEA5C-001; C5831001 (Other: Alias Study Number); 2023-505858-18-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-11-09; First posted 2023-11-14 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung; Stomach Neoplasms; Pancreatic Ductal Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma; Small Cell Lung Carcinoma
Keywords: CRC; NSCLC; PDAC; GC; GEJ; SCLC; Seattle Genetics
MeSH Terms: conditions — Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung; Stomach Neoplasms; Small Cell Lung Carcinoma | interventions — Bevacizumab; Fluorouracil; Oxaliplatin; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- PF-08046050 (Experimental): PF-08046050 monotherapy
  Interventions: Drug: PF-08046050
- PF-08046050 +bevacizumab (Experimental): PF-08046050 combination with bevacizumab
  Interventions: Drug: PF-08046050; Drug: bevacizumab
- PF-08046050 + bevacizumab + 5FU/LV (Experimental): PF-08046050 combination with bevacizumab + 5FU/LV
  Interventions: Drug: PF-08046050; Drug: bevacizumab; Drug: 5-Fluorouracil (5-FU); Drug: Leucovorin (LV)
- PF-08046050 + 5FU/LV + oxaliplatin + bevacizumab (Experimental): PF-08046050 combination with 5FU/LV + oxaliplatin + bevacizumab
  Interventions: Drug: PF-08046050; Drug: bevacizumab; Drug: 5-Fluorouracil (5-FU); Drug: Oxaliplatin; Drug: Leucovorin (LV)
- PF-08046050 + 5FU/LV + oxaliplatin (Experimental): PF-08046050 combination with 5FU/LV + oxaliplatin
  Interventions: Drug: PF-08046050; Drug: 5-Fluorouracil (5-FU); Drug: Oxaliplatin; Drug: Leucovorin (LV)
- PF-08046050 + 5FU/LV (Experimental): PF-08046050 combination with 5FU/LV
  Interventions: Drug: PF-08046050; Drug: 5-Fluorouracil (5-FU); Drug: Leucovorin (LV)

INTERVENTIONS:
Drug: PF-08046050 — Given into the vein (IV; intravenous)
  Other Names: SAR445953; SGN-CEACAM5C
Drug: bevacizumab — Given into the vein (IV; intravenous)
  Arms: PF-08046050 + 5FU/LV + oxaliplatin + bevacizumab; PF-08046050 + bevacizumab + 5FU/LV; PF-08046050 +bevacizumab
Drug: 5-Fluorouracil (5-FU) — Given into the vein (IV; intravenous)
  Arms: PF-08046050 + 5FU/LV; PF-08046050 + 5FU/LV + oxaliplatin; PF-08046050 + 5FU/LV + oxaliplatin + bevacizumab; PF-08046050 + bevacizumab + 5FU/LV
Drug: Oxaliplatin — Given into the vein (IV; intravenous)
  Arms: PF-08046050 + 5FU/LV + oxaliplatin; PF-08046050 + 5FU/LV + oxaliplatin + bevacizumab
Drug: Leucovorin (LV) — Given into the vein (IV; intravenous)
  Arms: PF-08046050 + 5FU/LV; PF-08046050 + 5FU/LV + oxaliplatin; PF-08046050 + 5FU/LV + oxaliplatin + bevacizumab; PF-08046050 + bevacizumab + 5FU/LV

SUMMARY:
This clinical trial is studying advanced solid tumors. Solid tumors are cancers that start in a part of your body like your lungs or liver instead of your blood. Once tumors have grown bigger in one place but haven't spread, they're called locally advanced. If your cancer has spread to other parts of your body, it's called metastatic. When a cancer has gotten so big it can't easily be removed or has spread to other parts of the body, it is called unresectable. These types of cancer are harder to treat.

Participants in this study must have cancer that has come back or did not get better with treatment. Participants must have a solid tumor cancer that can't be treated with standard of care drugs.

This clinical trial uses an experimental drug called PF-08046050. PF-08046050 is a type of antibody-drug conjugate or ADC. ADCs are designed to stick to cancer cells and kill them. They may also stick to some normal cells.

This study will test the safety of PF-08046050 in participants with solid tumors that are hard to treat or have spread throughout the body.

This study has 5 different study parts. Part A and Part B of the study will find out how much PF-08046050 should be given to participants. Part C will use the information from Parts A and B to see if PF-08046050 is safe and if it works to treat certain solid tumor cancers. Part D and E of the study, together with information from Parts A and B, will find out how much PF-08046050 should be given in combination with other anti-cancer agents. Part E will use the information from Parts A, B, and D to see if PF-08046050 is safe in combination with other anti-cancer agents and if it works to treat a certain solid tumor.

ELIGIBILITY:
Inclusion Criteria:

1. Tumor type:

   * Participants in Part A (dose escalation) and Part B (dose optimization) must have histologically- or cytologically-confirmed metastatic or unresectable solid tumor malignancy. Must have relapsed, refractory, or progressive disease, and should have no appropriate standard therapy available.

     * Participants in Part A must have one of the following tumor types: colorectal cancer (CRC); gastric carcinoma (GC) or gastroesophageal junction adenocarcinoma (GEJ); non-small cell lung cancer (NSCLC); or pancreatic ductal adenocarcinoma (PDAC).
     * The tumor types to be enrolled in Part B will be identified by the sponsor from among those specified in Part A.
   * Participants in Part C (dose expansion) must have one of the following histologically- or cytologically-confirmed metastatic or unresectable solid tumor malignancies.

     * CRC (adenocarcinoma of the colon or rectum) and must have received no more than 2 prior chemotherapy regimens for the treatment of advanced colorectal cancer and evidence of either progressive disease or intolerance to their last regimen.
     * PDAC with one or more metastatic lesions measurable by computed tomography/magnetic resonance imaging according to RECIST v1.1 criteria; and must have received no more than 1 prior chemotherapy regimen for the treatment of advanced PDAC and evidence of either progressive disease or intolerance to that regimen.
     * GC or GEJ and must have received prior platinum and fluoropyrimidine-based chemotherapy.
     * NSCLC and must have received platinum-based therapy. If eligible and consistent with local standard of care must have received a PD-1/PD-L1 inhibitor. In addition, participants with tumor genomic mutations/alterations for which approved targeted therapies are available per local standard of care, must have received such therapies.
     * Small cell lung cancer (SCLC) and must have received platinum-based therapy for extensive-stage disease and no more than 3 prior lines of therapy. If eligible and consistent with local standard of care must have received a PD 1/PD-L1 inhibitor.
   * CRC participants in Part D and Part E (bevacizumab combination therapy) must have histologically confirmed unresectable or metastatic adenocarcinoma of the colon or rectum. Received a maximum of 2 prior chemotherapy regimens for the treatment of advanced colorectal cancer and had demonstrated progressive disease or intolerance to their last regimen.
   * CRC participants in Part D and Part E (5FU/LV + bevacizumab and 5FU/LV + oxaliplatin + bevacizumab combination therapy) must have histologically confirmed unresectable or metastatic adenocarcinoma of the colon or rectum. Must not have received a prior TOPO1 inhibitor (such as irinotecan or nanoliposomal irinotecan) in any setting. 1L cohorts: No prior chemotherapy for advanced disease. 2L cohorts (applicable to 5FU/LV + bevacizumab combination only): 1 prior chemotherapy regimen for the treatment of advanced disease, which must have included a fluoropyrimidine and oxaliplatin.

   > 2L PDAC participants in Part E (5FU/LV combination therapy) must have histologically or cytologically confirmed metastatic pancreatic ductal adenocarcinoma. One or more metastatic lesions measurable by computed tomography/magnetic resonance imaging according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria.

   > 1L PDAC participants in Part E (5FU/LV + oxaliplatin combination therapy) must have histologically or cytologically confirmed metastatic pancreatic ductal adenocarcinoma that has not been previously treated in the metastatic setting. One or more metastatic lesions measurable by computed tomography/magnetic resonance imaging according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria. No prior chemotherapy for PDAC with the following exception: Patients who received adjuvant/neoadjuvant chemotherapy and who had recurrence more than 12 months after completion of adjuvant/neoadjuvant chemotherapy are eligible.
2. Participants enrolled in the following study parts should have a tumor site that is accessible for biopsy(ies) and agree to biopsy(ies) and/or submission of archival tissue:

   * Monotherapy dose optimization (Part B)
   * Monotherapy (Part C) and combination therapy (Part E) disease-specific expansion cohorts
3. An Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1
4. Measurable disease per Response Evaluation in Solid Tumors (RECIST) v1.1 at baseline.

Exclusion Criteria:

1. Previous exposure to CEACAM5-targeted therapy.
2. Prior treatment with a TOPO1-targeting ADC (CPT payload), such as Enhertu (trastuzumab deruxtecan) or Trodelvy (sacituzumab govitecan).
3. History of another malignancy within 3 years before the first dose of study intervention, or any evidence of residual disease from a previously diagnosed malignancy.
4. Active cerebral/meningeal disease related to the underlying malignancy. Participants with a history of cerebral/meningeal disease related to the underlying malignancy are allowed if prior central nervous system disease has been treated and the participant is clinically stable (defined as not having received steroid treatment for symptoms related to cerebral/meningeal disease for at least 2 weeks prior to enrollment and with no ongoing related AEs).

   > Criteria related to bevacizumab administration (participants in Parts D and E)
5. History of allergic reactions or hypersensitivity to bevacizumab or any of its excipients.
6. History of hypersensitivity to Chinese Hamster Ovary cell products or other recombinant human or humanized antibodies.
7. Serious non-healing wound, non-healing ulcer, or non-healing bone fracture.
8. Deep venous thromboembolic event within 4 weeks prior to enrollment
9. Known coagulopathy that increases risk of bleeding, bleeding diatheses.
10. History of any life-threatening VEGF-related adverse event

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 914 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2029-09-12 (Estimated); Study Completion 2030-09-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Through 30-37 days after the last study treatment, up to approximately 2 years
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention
Number of participants with laboratory abnormalities | Through 30-37 days after the last study treatment, up to approximately 2 years
Number of dose modifications due to AEs | Through end of treatment up to approximately 2 years
Number of participants with dose-limiting toxicities (DLTs) | Up to 28 days
Number of participants with DLTs by dose level | Up to 28 days

SECONDARY OUTCOMES:
Pharmacokinetic (PK) parameter - Area under the concentration-time curve (AUC) | Through 30-37 days after the last study treatment, up to approximately 2 years
  PK endpoint
PK parameter - Maximum concentration (Cmax) | Through 30-37 days after the last study treatment, up to approximately 2 years
  PK endpoint
PK parameter - Time to maximum concentration (Tmax) | Through 30-37 days after the last study treatment, up to approximately 2 years
  PK endpoint
PK parameter - Trough concentration (Ctrough) | Through 30-37 days after the last study treatment, up to approximately 2 years
  PK endpoint
Number of participants with antidrug antibodies (ADAs) | Through 30-37 days after the last study treatment, up to approximately 2 years
Objective response rate (ORR) | Through end of study and up to approximately 2 years
  The objective response rate (ORR) is defined as the percentage of participants with complete response (CR) or partial response (PR) which is subsequently confirmed as assessed according to Response Evaluation in Solid Tumors (RECIST) v1.1.
Best overall response | Through end of study and up to approximately 2 years
  The best overall response for a participant will be determined by the order of confirmed CR, confirmed PR, stable disease (SD), progressive disease (PD), not evaluable (NE) or not applicable (NA) per RECIST v1.1.
Duration of response (DOR) | Through end of study and up to approximately 2 years
  DOR is defined as the time from start of the first documentation of objective tumor response (CR or PR) to the first documentation of tumor progression per RECIST v1.1 or to death due to any cause
Progression-free survival (PFS) | Through end of study and up to approximately 2 years
  PFS is defined as the time from start of SGN-CEACAM5C to first documentation of disease progression (based on radiographic assessments per RECIST v1.1) or death due to any cause, whichever comes first
Overall survival (OS) | Through end of study and up to approximately 2 years
  OS is defined as the time from start of SGN-CEACAM5C to date of death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (43):
- United States (21):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Mayo Clinic, Scottsdale, Arizona
  - City of Hope (City of Hope National Medical Center, City of Hope Medical Center), Duarte, California
  - IP Address: City of Hope Investigational Drug Services(IDS), Duarte, California
  - University of Colorado Hospital - Anschutz Cancer Pavilion (ACP), Aurora, Colorado
  - University of Colorado Hospital/University of Colorado, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - Florida Cancer Specialists, Orlando, Florida
  - Sarah Cannon Research Institute at Florida Cancer Specialists, Orlando, Florida
  - School of Medicine, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer at Johns Hopkins, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - START Midwest, Grand Rapids, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Sarah Cannon Research Institute - Pharmacy, Nashville, Tennessee
  - SCRI Oncology Partners, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - South Texas Accelerated Research Therapeutics, LLC, San Antonio, Texas
  - START Mountain Region, Salt Lake City, Utah
  - South Texas Accelerated Research Therapeutics Mountain Region, West Valley City, Utah
- Canada (5):
  - The Ottawa Hospital, Ottawa, Ontario
  - University Health Network, Toronto, Ontario
  - University Health Network, Princess Margaret Cancer Centre, Toronto, Ontario
  - The Research Institute of the McGill University Health Centre, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
- France (2):
  - Institut Gustave Roussy, Villejuif, Paris
  - Gustave Roussy, Villejuif
- Netherlands Cancer Institute, Amsterdam, Netherlands
- Spain (5):
  - Institut Catala d'Oncologia - Hospital Duran i Reynals (ICO L'Hospitalet), L'Hospitalet de Llobregat, Catalunya [cataluña]
  - Ascires Cetir, Barcelona
  - Ascires CETIR, Esplugues de Llobregat
  - Servicio de Farmacia ICO - Planta 0, L'Hospitalet de Llobregat
  - Hospital Universitario HM Sanchinarro-CIOCC-START Madrid, Madrid
- Sweden (2):
  - Karolinska University Hospital, Solna
  - ApoEx NKS, Stockholm
- United Kingdom (7):
  - Diagnostic Centre, London, Others
  - The Harley Street Clinic (THSC), London, Other
  - Edinburgh Cancer Centre, Western General Hospital, Edinburgh, Scotland
  - Western General Hospital, Edinburgh
  - Sarah Cannon Research Institute UK, London
  - The Harley Street Clinic, London
  - Radiology, London

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=SGNCEA5C-001